CLINICAL TRIAL: NCT07200180
Title: Perioperative Argon Inhalation to Improve Neurocognitive Recovery After Carotid Surgery (PAIRS Trial)
Brief Title: Perioperative Argon Inhalation to Improve Neurocognitive Recovery After Carotid Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Negovsky Reanimatology Research Institute (Other Government)
Responsible Party: Principal Investigator, Oleg A. Grebenchikov, The head of the laboratory in the Negovsky Reanimatology Research Institute, Negovsky Reanimatology Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PAIRS
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Carotid Artery Disease; Carotid Artery Stenoses
Keywords: Carotid artery disease; Carotid artery stenosis; Carotid artery surgery; Neurocognitive disorders; postoperative delirium; Stroke; Neuroinflammation; Argon; Organ protection
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis; Neurocognitive Disorders; Emergence Delirium; Stroke; Neuroinflammatory Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Аrgon-oxygen breathing mixture (Experimental): Perioperative inhalation of an argon-oxygen mixture (70% argon, 30% oxygen)
  Interventions: Drug: Аrgon-oxygen breathing mixture
- Nitrogen-oxygen breathing mixture (Sham Comparator): Perioperative inhalation of an nitrogen-oxygen mixture (70% nitrogen, 30% oxygen)
  Interventions: Drug: Nitrogen-oxygen breathing mixture

INTERVENTIONS:
Drug: Аrgon-oxygen breathing mixture — Patients receive a course of inhalations with an argon-oxygen mixture according to the following protocol: 60 minutes on day 1 prior to surgery, 60 minutes one hour before being transferred to the operating room, and 60 minutes on the first postoperative day
  Arms: Аrgon-oxygen breathing mixture
Drug: Nitrogen-oxygen breathing mixture — Patients receive a course of inhalations with an nitrogen-oxygen mixture according to the following protocol: 60 minutes on day 1 prior to surgery, 60 minutes one hour before being transferred to the operating room, and 60 minutes on the first postoperative day
  Arms: Nitrogen-oxygen breathing mixture

SUMMARY:
Currently, over 400,000 reconstructive surgeries on carotid arteries are performed annually worldwide, including carotid endarterectomy (CEA) and carotid stenting. These interventions have proven effective in preventing ischemic stroke in patients with hemodynamically significant carotid artery stenoses. However, even following a technically successful procedure, the risk of perioperative ischemic brain injury persists. According to meta-analyses, one in five patients exhibits covert ("silent") strokes after reconstructive interventions, with their frequency being ten times higher than that of clinically manifest events. Such lesions are associated with cognitive decline and an increased risk of dementia. An additional risk factor is the "no-reflow" phenomenon-an impairment of microcirculatory reperfusion that occurs even after the restoration of macrovascular blood flow, thereby limiting the effectiveness of surgical revascularization.

Cognitive disorders and postoperative delirium, observed in 15-30% of patients after CEA, adversely affect rehabilitation and long-term prognosis. To date, there are no reliable pharmacological strategies to prevent these complications.

In this context, inert gases have attracted significant interest as potential neuroprotective agents. Xenon, despite its proven efficacy, is limited by high cost and challenges in industrial production. Argon, in contrast, is accessible, safe, and technologically straightforward to administer. In preclinical models of stroke and ischemia-reperfusion, argon has demonstrated pronounced anti-apoptotic, anti-inflammatory, and antioxidant effects, mediated through the regulation of TLR2/4-, ERK1/2-, Nrf2-, and NF-κB-dependent signaling pathways. Its ability to suppress microglial activation towards the M1 phenotype and inhibit the NLRP3 inflammasome has been noted, which reduces neuroinflammation and decreases the volume of secondary neuronal damage. Short-term argon inhalation in healthy volunteers has shown a favorable safety profile with no adverse effects on cerebral hemodynamics.

Thus, it is highly relevant to clinically test the hypothesis that perioperative inhalation of an argon-containing gas mixture can reduce the incidence of ischemic brain injuries and cognitive impairments in patients undergoing CEA.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* elective carotid artery surgery
* general anesthesia
* written informed consent

Exclusion Criteria:

* The presence of any mental disorder according to the International Classification of Diseases 10th Revision which is confirmed by a psychiatrist.
* The presence of any neuromuscular disease according to the International Classification of Diseases 10th Revision
* Heart failure equal 3 or 4 class according to the New York Heart Association Functional Classification
* Pregnant or breast-feeding women
* Inability to undergo a preoperative assessment for any reason
* Previously enrolled in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | 30 days
  Number of patients with even one positive confusion assessment method for the intensive care unit or 3-minute confusion assessment method

SECONDARY OUTCOMES:
Incidence of emergence delirium | 30 days
  Number of patients with positive the confusion assessment method for the intensive care unit as soon as they reach Aldrete score of 9 points
Incidence of postoperative agitation | 30 days
  Richmond agitation-sedation scale more or equal +2 evaluated from the end of volatile anesthetic supply to the moment when a patient reaches Aldrete score of 9 points Richmond agitation-sedation scale: minimum value = -5 (Unarousable - no response to voice or physical stimulation) maximum value = +4 (Combative - overtly combative or violent; immediate danger to staff) Adequate patients have the results of Richmond agitation-sedation score equal 0 (Alert and calm; Spontaneously pays attention to caregiver)
Duration of postoperative delirium | until 1 month after surgery
  30 days - number of days in which patient had positive confusion assessment method for the intensive care unit or 3-minute confusion assessment method
Incidence of cognitive dysfunction | 30 days
  reduction of ≥1 standard deviation in the Montreal Cognitive Assessment (MoCA) total z-score compared to the preoperative assessment
Incidence of overt stroke | 30 days
  Number of overt strokes
Incidence of covert stroke | 30 days
  Number of covert strokes
Length of stay in the intensive care unit | 30 days
  Number of days in intensive care unit
Length of hospitalization | 30 days
  Number of days in hospital
Serum level of S100 beta protein | 2 days after surgery
  Serum level of S100 beta protein
Serum level of neuron-specific enolase | 2 days after surgery
  Serum level of neuron-specific enolase
Serum level of interleukin-6 | 2 days after surgery
  Serum level of interleukin-6

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Grebenchikov, MD, PhD, Principal Investigator — Negovsky Reanimatology Research Institute
Locations (1):
- Demikhov Municipal Clinical Hospital 68, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Decision of the local ethics committee